CLINICAL TRIAL: NCT05632042
Title: Response of Metabolic Syndrome and Sexual Dysfunction to Lifestyle Changes/Modifications in Men With Psoriasis
Brief Title: Response of Metabolic Syndrome and Sexual Dysfunction to Lifestyle Changes in Men With Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004117
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Psoriasis; Metabolic Syndrome; Erectile Dysfunction
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome; Erectile Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle-modification group (Experimental): erectile dysfunction (ED) psoriatic men with metabolic syndrome (group = 30 patients) will receive lifestyle changes (12 weeks of low calorie diet and moderate-intensity walking on treadmill, the walking duration will be 40 minutes, the walking will be three times per week)
  Interventions: Behavioral: lifestyle modification (exercise and control of diet)
- control group (No Intervention): erectile dysfunction (ED) psoriatic men with metabolic syndrome (number of the patients will be 30) that will receive no lifestyle changes/modifications.

INTERVENTIONS:
Behavioral: lifestyle modification (exercise and control of diet) — erectile dysfunction (ED) psoriatic men with metabolic syndrome that will receive lifestyle changes (12 weeks of low calorie diet and moderate-intensity walking on treadmill, the walking duration will be 40 minutes, the walking will be three times per week)
  Arms: lifestyle-modification group

SUMMARY:
complaint of sexual dysfunction and metabolic syndrome are highly reported in men with psoriasis

DETAILED DESCRIPTION:
erectile dysfunction (ED) psoriatic men with metabolic syndrome (number of the patients will be 60) will assigned to study group (group = 30 patients) that will receive lifestyle changes (12 weeks of low calorie diet and moderate-intensity walking on treadmill, the walking duration will be 40 minutes, the walking will be three times per week) or control group (group=30 patients) that will receive no lifestyle changes/modifications.

ELIGIBILITY:
Inclusion Criteria:

* psoriatic married men with metabolic syndrome and erectile dysfunction

Exclusion Criteria:

* patients with heart, respiratory, other autoimmune problems

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity
Enrollment: 60 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-04-16 (Estimated); Study Completion 2023-04-16 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function | It will be measured after 12-week intervention
  Arabic version of this 5-item questionnaire will used to assess erectile function/dysfunction

SECONDARY OUTCOMES:
psoriasis area and severity index | It will be measured after 12-week intervention
  it is a tool used to measure the severity and extent of psoriasis.
body mass index | It will be measured after 12-week intervention
  patients will be assessed with empty bowel and bladder
systolic blood pressure | It will be measured after 12-week intervention
  it will be measured using sphygmomanometer
diastolic blood presure | It will be measured after 12-week intervention
  it will be measured using sphygmomanometer
waist circumference | It will be measured after 12-week intervention
  it will be measured by in elastic tape
blood glucose | It will be measured after 12-week intervention
  it will be measured in fasting status
triglycerides | It will be measured after 12-week intervention
  it will be measured in serum
high density lipoprotein | It will be measured after 12-week intervention
  it will be measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt